CLINICAL TRIAL: NCT03030859
Title: Self-Care for Head and Neck Cancer Survivors With Lymphedema and Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: American Cancer Society, Inc. (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jie Deng, Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB# 828744; NCI-2016-01901 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2016-12-30; First posted 2017-01-25 (Estimated); Results first posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Cancer; Lymphedema; Fibrosis
MeSH Terms: conditions — Head and Neck Neoplasms; Lymphedema; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Usual Care) (Experimental): Patients receive usual care only, without any additional interventions.
  Interventions: Other: Usual Care
- Group II (Usual Care plus LEF-SCP) (Experimental): Patients undergo LEF-SCP training comprising of MI session over 1 hour and LEF self-care training session over 1 hour weekly for 3 weeks. Patients also review LEF self-care educational manual and watch self-care videos monthly or more frequently as needed.
  Interventions: Other: Usual Care plus LEF-SCP
- Group III (Usual Care plus LEF-SCP plus Follow-Up) (Experimental): Patients undergo LEF-SCP training comprising of MI session over 1 hour and LEF self-care training session over 1 hour weekly for 3 weeks. Patients review LEF self-care educational manual and watch self-care videos monthly or more frequently as needed. Patients also meet with the study lymphedema therapist over 1 hour at 3, 6, and 9 months.
  Interventions: Other: Usual Care plus LEF-SCP plus Follow-up

INTERVENTIONS:
Other: Usual Care — Undergo usual care only
  Arms: Group I (Usual Care)
Other: Usual Care plus LEF-SCP — Undergo Motivational Interviewing sessions and LEF Self-Care Training sessions, as well as review LEF self-care educational manual and videos
  Arms: Group II (Usual Care plus LEF-SCP)
Other: Usual Care plus LEF-SCP plus Follow-up — Undergo Motivational Interviewing sessions and LEF Self-Care Training sessions, and review LEF self-care educational manual and videos, as well as meet with the study lymphedema therapist
  Arms: Group III (Usual Care plus LEF-SCP plus Follow-Up)

SUMMARY:
This randomized pilot clinical trial studies how well the self-care program works in head and neck cancer survivors with lymphedema and fibrosis. A self-care program may promote self-care activities for managing chronic swelling and tough/tight tissues in the head and neck region.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To complete development of a self-care program focusing on lymphedema and fibrosis (LEF) in head and neck cancer (HNC) survivors (LEF-self-care program [SCP]) with the goal of improving LEF associated outcomes when compared to usual care alone. (Stage I)

II. To determine the feasibility of a program of LEF-SCP with or without follow-up to usual care for HNC survivors with LEF, specifically to: 1) obtain recruitment estimates and determine barriers to recruitment; 2) identify barriers to implementation; 3) assess safety; and 4) evaluate patient satisfaction. (Stage II)

III. To determine if the LEF-SCP with or without follow-up enhances self-efficacy and adherence compared to usual care in HNC survivors with LEF. (Stage II)

IV. To determine the preliminary efficacy of the LEF-SCP with or without follow-up as compared to usual care for the following outcomes: 1) LEF progression; 2) symptom burden; and 3) functional status. (Stage II)

OUTLINE:

Project Stage I: Patients undergo a training session with the study lymphedema therapist and review the educational manual and videos for the development of all three components of the LEF self-care program.

Project Stage II: Patients are randomized to 1 of 3 groups.

GROUP I: Patients will receive usual care only, without any additional interventions.

GROUP II: Patients undergo LEF-SCP training comprising of motivational interview (MI) session over 1 hour and LEF self-care training session over 1 hour weekly for 3 weeks. Patients also review LEF self-care educational manual and watch self-care videos monthly or more frequently as needed.

GROUP III: Patients undergo LEF-SCP training comprising of MI session over 1 hour and LEF self-care training session over 1 hour weekly for 3 weeks. Patients review LEF self-care educational manual and watch self-care videos monthly or more frequently as needed. Patients also meet with the study lymphedema therapist over 1 hour at 3, 6, and 9 months.

After completion of study, patients are followed up at 3, 6, 9, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Post HNC primary treatment
* No evidence of cancer (NED)
* No more than 6 months after completion of initial lymphedema therapy for head and neck lymphedema
* > 18 years of age
* Ability to understand English in order to complete questionnaires
* Able to complete the onsite training and home self-care activities for LEF management
* Able to provide informed consent

Exclusion Criteria:

• Patients will be excluded if they have any of the following medical conditions that would prohibit the safe implementation of self-care of LEF: recurrent or metastatic cancer; any other active cancer; acute infection; congestive heart failure; renal failure; cardiac or pulmonary edema; sensitive carotid sinus; severe carotid blockage; and uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jie Deng, PhD, RN, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Deng J, Murphy BA, Andersen LP, McMenamin E, Lukens JN, Cohn JC, Rajasekaran K, Quinn RJ, Spinelli BA, Lin A. Feasibility and preliminary efficacy of a lymphedema and fibrosis self-management program for head and neck cancer survivors: a pilot randomized controlled trial. Oral Oncol. 2025 Sep;168:107556. doi: 10.1016/j.oraloncology.2025.107556. Epub 2025 Aug 6. PMID 40773982
- [Derived] Deng J, Lukens JN, Cohn JC, McMenamin E, Murphy B, Spinelli BA, Murphy N, Steinmetz AK, Landriau MA, Lin A. Conducting a supportive oncology clinical trial during the COVID-19 pandemic: challenges and strategies. Trials. 2022 Nov 8;23(1):927. doi: 10.1186/s13063-022-06804-w. PMID 36348346
- [Derived] Deng J, Dietrich MS, Murphy B. Self-care for head and neck cancer survivors with lymphedema and fibrosis: study protocol for a randomized controlled trial. Trials. 2019 Dec 27;20(1):775. doi: 10.1186/s13063-019-3819-0. PMID 31882012

RESULTS

PARTICIPANT FLOW:
Groups:
- Group I (Usual Care): Participants received usual care.
- Group II (Usual Care Plus LEF-SM Program): Participants received usual care and LEF-SM Program.
- Group III (Usual Care Plus LEF-SM Program Plus Follow-Up With a Lymphedema Therapist): Participants received usual care plus LEF-SM Program plus follow-up with a lymphedema therapist
Period: Overall Study
Arm/Group | Group I (Usual Care) | Group II (Usual Care Plus LEF-SM Program) | Group III (Usual Care Plus LEF-SM Program Plus Follow-Up With a Lymphedema Therapist)
Started | 20 | 20 | 19
Completed | 19 | 17 | 13
Not Completed | 1 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Group I (Usual Care): Patients receive monthly automated system telephone call for 12 months.
  Usual Care: Undergo usual care only
- Group II (Usual Care Plus LEF-SCP): Patients undergo LEF-SCP training comprising of MI session over 1 hour and LEF self-care training session over 1 hour weekly for 3 weeks. Patients receive monthly automated system telephone call for 12 months. Patients also review LEF self-care educational manual and watch self-care videos monthly or more frequently as needed.
  Usual Care plus LEF-SCP: Undergo Motivational Interviewing sessions and LEF Self-Care Training sessions, as well as review LEF self-care educational manual and videos
- Group III (Usual Care Plus LEF-SCP Plus Follow-Up): Patients undergo LEF-SCP training comprising of MI session over 1 hour and LEF self-care training session over 1 hour weekly for 3 weeks. Patients receive monthly automated system telephone call for 12 months. Patients review LEF self-care educational manual and watch self-care videos monthly or more frequently as needed. Patients also meet with the study lymphedema therapist over 1 hour at 3, 6, and 9 months.
  Usual Care plus LEF-SCP plus Follow-up: Undergo Motivational Interviewing sessions and LEF Self-Care Training sessions, and review LEF self-care educational manual and videos, as well as meet with the study lymphedema therapist
- Total: Total of all reporting groups
Arm/Group | Group I (Usual Care) | Group II (Usual Care Plus LEF-SCP) | Group III (Usual Care Plus LEF-SCP Plus Follow-Up) | Total
Number analyzed (Participants) | 20 | 20 | 19 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (7.5) | 60 (10.9) | 60 (11.0) | 60 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 2 | 10
  Male | 16 | 16 | 17 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 4 | 1 | 5
  White | 20 | 15 | 18 | 53
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 19 | 59

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the LEF-SCP (Self-Care Skill Training Sessions)
Description: Feasibility of the LEF-SCP was evaluated by number of participants that completed the self-care skill training sessions (at least 2 out of 3 sessions). This measure was applicable to Group II and Group III only.
Time Frame: Following 3 weeks of the LEF-SCP sessions
Measure: Count of Participants; unit: Participants
Arm/Group | Group II (Usual Care Plus LEF-SCP) | Group III (Usual Care Plus LEF-SCP Plus Follow-Up)
Number analyzed (Participants) | 20 | 19
Participants | 20 | 18

2. Primary Outcome: Feasibility of the LEF-SCP (Motivational Interviewing Sessions)
Description: Feasibility of the LEF-SCP was evaluated by number of participants that completed the motivational interviewing sessions (at least 2 out of 3 sessions). This measure was applicable to Group II and Group III only.
Time Frame: Following 3 weeks of motivational interviewing sessions
Measure: Count of Participants; unit: Participants
Arm/Group | Group II (Usual Care Plus LEF-SCP) | Group III (Usual Care Plus LEF-SCP Plus Follow-Up)
Number analyzed (Participants) | 20 | 18
Participants | 20 | 16

3. Primary Outcome: Preliminary Efficacy of the LEF-SCP (Total Severity of External LEF)
Description: Change in total severity of external LEF from baseline to 12 months post-intervention. A larger change in this score means more reduction in the severity of external LEF,
  External LEF is measured by HN-LEF Assessment Criteria. The total external LEF severity score is calculated by summing the severity score of each site (total 9 sites, severity score ranging from 0-27). For each site, the severity of LEF includes no LEF (=0), mild (=1), moderate (=2), and severe (=3).
Time Frame: at 12 months post-intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Group 1: Usual Care
- Group 2: Usual Care Plus LEF-SCP
- Group 3: Usual Care Plus LEF-SCP Plus Follow-Up
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 19 | 20 | 16
score on a scale | -0.11 [-1.01 to 0.80] | -2.35 [-3.51 to -1.19] | -2.25 [-3.91 to -0.59]

4. Primary Outcome: Preliminary Efficacy of the LEF-SCP (Symptom Burden)
Description: Change in symptom burden score from baseline to 12 months post-intervention. A larger change in this score means decreased symptom burden.
  Symptom burden is assessed by Head and Neck Lymphedema and Fibrosis Symptom Inventory (HN-LEF SI). Higher scores (score ranging from 0-5) indicate increased symptom burden. There are 7 subscales and only one subscale (soft tissue and neurologic toxicity) score is reported here.
Time Frame: at 12 months post-intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 19 | 20 | 16
score on a scale | -0.15 [-0.49 to 0.19] | -0.73 [-1.21 to -0.24] | -0.53 [-1.06 to -0.01]

5. Primary Outcome: Preliminary Efficacy of the LEF-SCP (Self-Efficacy)
Description: Change in self-efficacy score from baseline to 12 months post-intervention. A larger change in this score means increased self-efficacy.
  Self-efficacy is assessed by Perceived Medical Condition Self-Management Scale (PMCSMS) (8-item). Higher scores (score ranging from 8-40) indicate greater self-efficacy.
Time Frame: at 12 months post-intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 19 | 17 | 13
score on a scale | 1.26 [-1.33 to 3.85] | 4.71 [1.21 to 8.21] | 4.85 [0.12 to 9.57]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 12 months.
Description: No adverse event was reported during the study.
Arm/Group | Group I (Usual Care) | Group II (Usual Care Plus LEF-SCP) | Group III (Usual Care Plus LEF-SCP Plus Follow-Up)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/19

LIMITATIONS AND CAVEATS:
This was a pilot study with the small number of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/59/NCT03030859/Prot_SAP_000.pdf